CLINICAL TRIAL: NCT01823887
Title: Autonomic Neural Regulation Therapy to Enhance Myocardial Function in Heart Failure (ANTHEM-HF) Study
Acronym: ANTHEM-HF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-01
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; Vagus Nerve; VNS
MeSH Terms: conditions — Heart Failure | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left Sided Stimulation (Experimental): Left cervical Vagus Nerve Stimulation (VNS)
  Interventions: Device: Vagus Nerve Stimulation (VNS)
- Right Sided Stimulation (Experimental): Right Cervical Vagus Nerve Stimulation (VNS)
  Interventions: Device: Vagus Nerve Stimulation (VNS)

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) — Electrical Stimulation of the Vagus Nerve

SUMMARY:
The ANTHEM-HF Study is designed to demonstrate the safety and efficacy of vagus nerve stimulation (VNS) with the Cyberonics VNS Therapy System for the treatment of subjects with symptomatic heart failure.

DETAILED DESCRIPTION:
Heart failure patients will be enrolled and randomized to cervical VNS implantation on either the left side or right side. After a 2-week post-implantation recovery period and a 10-week stimulation titration period, continuous periodic stimulation will be performed for 6 months, with data collection at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic heart failure, New York Heart Association (NYHA) class II/III with reduced EF and dilated hearts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cardiac Function | 6 months
  Left ventricular end-systolic volume (LVESV) and ejection fraction (EF)
Adverse Events | 6 months
  Incidence of procedure and device-related complications

SECONDARY OUTCOMES:
Functional Status | 6 months
  6-minute walk test
Quality of Life | 6 months
  Minnesota Living with Heart Failure Questionnaire
Functional Status | 6 months
  New York Heart Association Class
Autonomic Function | 6 months
  Heart Rate Variability (HRV)
Blood Biomarkers | 6 months
  Blood Levels of Heart Failure Biomarkers
Cardiac Function | 6 months
  Left ventricular end-systolic diameter (LVESD)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Cyberonics, Inc.
Locations (1):
- Chennai, India

REFERENCES:
- [Background] Dicarlo L, Libbus I, Amurthur B, Kenknight BH, Anand IS. Autonomic regulation therapy for the improvement of left ventricular function and heart failure symptoms: the ANTHEM-HF study. J Card Fail. 2013 Sep;19(9):655-60. doi: 10.1016/j.cardfail.2013.07.002. PMID 24054343
- [Result] Premchand RK, Sharma K, Mittal S, Monteiro R, Dixit S, Libbus I, DiCarlo LA, Ardell JL, Rector TS, Amurthur B, KenKnight BH, Anand IS. Autonomic regulation therapy via left or right cervical vagus nerve stimulation in patients with chronic heart failure: results of the ANTHEM-HF trial. J Card Fail. 2014 Nov;20(11):808-16. doi: 10.1016/j.cardfail.2014.08.009. Epub 2014 Sep 1. PMID 25187002
- [Derived] Libbus I, Premchand RK, Sharma K, Mittal S, Monteiro R, Amurthur B, KenKnight BH, DiCarlo LA, Anand IS. Persistent Autonomic Engagement and Cardiac Control After Four or More Years of Autonomic Regulation Therapy Using Vagus Nerve Stimulation. Front Physiol. 2022 Mar 11;13:853617. doi: 10.3389/fphys.2022.853617. eCollection 2022. PMID 35360224
- [Derived] Nearing BD, Libbus I, Carlson GM, Amurthur B, KenKnight BH, Verrier RL. Chronic vagus nerve stimulation is associated with multi-year improvement in intrinsic heart rate recovery and left ventricular ejection fraction in ANTHEM-HF. Clin Auton Res. 2021 Jun;31(3):453-462. doi: 10.1007/s10286-021-00780-y. Epub 2021 Feb 16. PMID 33590355
- [Derived] Nearing BD, Libbus I, Amurthur B, Kenknight BH, Verrier RL. Acute Autonomic Engagement Assessed by Heart Rate Dynamics During Vagus Nerve Stimulation in Patients With Heart Failure in the ANTHEM-HF Trial. J Cardiovasc Electrophysiol. 2016 Sep;27(9):1072-7. doi: 10.1111/jce.13017. Epub 2016 Jul 7. PMID 27221316
- [Derived] Libbus I, Nearing BD, Amurthur B, KenKnight BH, Verrier RL. Autonomic regulation therapy suppresses quantitative T-wave alternans and improves baroreflex sensitivity in patients with heart failure enrolled in the ANTHEM-HF study. Heart Rhythm. 2016 Mar;13(3):721-8. doi: 10.1016/j.hrthm.2015.11.030. Epub 2015 Nov 18. PMID 26601770